CLINICAL TRIAL: NCT02136264
Title: Randomized Controlled Trial of a Personalized Dietary Intervention Approach for the Control of Essential Hypertension
Brief Title: Study of Personalized Dietary Intervention for the Control of Essential Hypertension
Acronym: PCFADASH-HT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nigeria, Enugu Campus (Other)
Collaborators: University of Glasgow (Other); University Of Nigeria Teaching Hospital (Network)
Responsible Party: Principal Investigator, Dr C.P. Chijioke, Professor C.P. Chijioke, University of Nigeria, Enugu Campus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PCFADASH-HT
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Essential Hypertension
Keywords: hypertension; dietary intervention; personalized nutrition; randomized controlled trial
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCFA interventional dietary counselling (Active Comparator): personalized categorical food avoidance dietary counselling
  Interventions: Other: PCFA interventional dietary counselling
- conventional DASH diet counselling (Sham Comparator): DASH = conventional "dietary approach to stop hypertension"
  Interventions: Other: conventional DASH diet counselling

INTERVENTIONS:
Other: PCFA interventional dietary counselling
  Arms: PCFA interventional dietary counselling
Other: conventional DASH diet counselling
  Arms: conventional DASH diet counselling

SUMMARY:
An ongoing case study of psoriasis, shows reproducibly that ingestion of hydrogenated fats, and some flavourant or sweetener compounds, leads to relapse of psoriasis, and secondary food intolerances, followed by remission over a couple of months (cpcpsoriasis.blogspot.com). Hence a personalized categorical food avoidance diet averts relapse and maintains remission of psoriasis, with side benefit on blood pressure and other metabolic parameters (J Hypertension 2012; 30: e-suppl 1, poster 158). Study hypothesis: this dietary approach would improve the control of essential hypertension. A randomized controlled clinical trial is proposed to compare this dietary approach with conventional DASH-type dietary counselling. 40 study participants will be randomly assigned to either conventional or interventional dietary counselling. They will be comprehensively monitored (including gene expression studies) for two years. Outcome criteria will include blood pressure, complications of hypertension, side-benefit on comorbidity, and requirement for antihypertensive drugs.

ELIGIBILITY:
Inclusion Criteria:

1. average blood pressure exceeds 160/100mm Hg (140/90 if additional vascular risk), regardless of whether on treatment
2. on one or two antihypertensive drugs AND average BP exceeds 140/90 (130/80 if additional risk)
3. on three or more antihypertensives, regardless of whether BP controlled
4. sufficiently literate to follow detailed dietary instructions
5. informed consent

Exclusion Criteria:

1. disabling complications of hypertension
2. secondary cause of hypertension
3. pregnancy
4. age less than 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
a statistically significant 12 mm Hg (or more) greater change of blood pressure in one group compared to the other | 2 years

SECONDARY OUTCOMES:
resolution of hypertension (normal blood pressure, no drugs required) | 2 years
serious (disabling) adverse events attributable to hypertension or its drug treatment | 2 years

OTHER OUTCOMES:
a reduction in antihypertensive treatment required i.e. reduced number of drugs required, or dosage of at least two drugs reduced by half | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chioli P Chijioke, MA MB BChir MD, Principal Investigator — College of Medicine, University of Nigeria
Locations (1):
- Chiolive International Medical Research Organisation, Enugu, Enugu State, Nigeria